CLINICAL TRIAL: NCT04470375
Title: Cohort Study of Use of Virtual Reality Pain Neuroscience Education for Middle School Students and Effects on Pain Knowledge and Beliefs
Brief Title: Virtual Reality Pain Neuroscience Education for Middle School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Kory Zimney, Associate Professor, University of South Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USD-IRB-20-129
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Pain; Education; Virtual Reality
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: single group of students receiving Virtual Reality education
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR pain education (Experimental): Students receiving the 45 minute pain education through Virtual Reality
  Interventions: Behavioral: Virtual Reality Pain Neuroscience Education

INTERVENTIONS:
Behavioral: Virtual Reality Pain Neuroscience Education — Use of virtual reality media to provide pain neuroscience education

SUMMARY:
Investigating the use of a Virtual Reality (VR) pain neuroscience education (PNE) platform with middle school students. The investigators have previously studied the use of PNE with in person educational sessions with middle school kids and video recorded sessions. This study will be looking into utilizing the VR platform for delivery of the educational information.

DETAILED DESCRIPTION:
Potential middle school students will be contacted through fliers to local parents in the Louisville, KY area via various sports team events. The investigators have secured a meeting room space at a large reception room at Lake Forest Country Club (Louisville, KY) on August 4, 2020. Potential participants will call to schedule time for participation to allow for proper staggering of participants arriving on the day of data collection.

Research team will set up informed consent space at the entrance to the reception room and stagger participant arrival time to reduce contact with other participants. This space will be cleaned and disinfected regularly during the consenting process as new participants arrive. Once student and parent arrives they will complete informed consent and COVID-19 screening form before being allowed into research space (reception room). Each participant will be given a pen to keep during the research study and go home with also provided with hand sanitizer to use before and after. No pens will be reused with other participants. Masks will be made available for anyone that requests one, but they will not be required while at the testing location. Parents of child will be allowed to sit in waiting chair keeping 6 feet of distance from anyone else. The child research participant will be lead to a chair in the room and complete pre-test questionnaire and then they will be set-up with a Virtual Reality (VR) device (cleaned and disinfected between each use) and go through a VR educational experience (~30 minutes) on Pain Neuroscience Education (PNE). Upon completion of the VR educational session they will complete post-test questionnaire and then be able to leave.

ELIGIBILITY:
Inclusion Criteria:

* willing to view VR educational session
* in grades 5, 6, 7, or 8.

Exclusion Criteria:

* has been through PNE educational program previously
* aversion to VR or problems with viewing VR in the past
* history of epilepsy or seizures
* eye surgery or injury within the last 6 months
* open sores or wounds around where VR googles are worn on face
* anyone who has had a concussion that has not been cleared for full activity or experiencing any post-concussion syndrome symptoms currently.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kory J Zimney, PT, DPT, Principal Investigator — University of South Dakota
Locations (1):
- Evidence in Motion (Lake Forest Country Clug), Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Data will be stored for required 3 year period after study. No intent at this time to share data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Middle school students (Grades 5-8), live in Louisville, KY area, no PNE training sessions in the past, no history of epilepsy or seizures or adverse events with viewing VR in the past.
Pre-assignment Details: No exclusion prior to assignment
Groups:
- Middle School VR Students: Middle school students viewing the VR on PNE
Period: Overall Study
Arm/Group | Middle School VR Students
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Middle school students
Arm/Group | Middle School VR Students
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.45 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
current pain [Count of Participants; unit: Participants]
  no | 19
  yes | 1
history of any previous pain [Count of Participants; unit: Participants]
  one week | 13
  one month | 4
  more than 3 months | 2
  Not reported | 1
Pain beliefs questionnaire [Mean (Standard Deviation); unit: scores on a scale] — Pain beliefs questions: answer on 11 point Likert Scale from strongly disagree=0 to strongly agree=10
  1. Pain is normal; without being able to feel pain you will not survive.
  2. Pain means something is wrong with your tissues
  3. Pain always means you have to stop what you are doing
  4. You can control how much pain you feel
  5. Your brain decides if you feel pain, not your tissues
  scores on a scale
    pain beliefs question 1. | 5.2 (3.1)
    pain beliefs question 2. | 4.1 (2.2)
    Pain beliefs question 3. | 1.95 (2.1)
    pain beliefs question 4. | 2.9 (3.1)
    pain beliefs question 5. | 5.7 (2.0)
revised Neurophysiology of Pain Questionnaire [Mean (Standard Deviation); unit: correct answers] — 12 true/false questions regarding the neurophysiology of pain. Answers of unsure are marked as incorrect answers as individuals are told not to guess at answer and only answer if they think they know the correct answer. Score is the number of correct answers provided.
  correct answers | 3.9 (1.6)
Physical activity Fear Avoidance Beliefs Questionnaire [Mean (Standard Deviation); unit: score on a scale] — Questionnaire on fear of physical activity. 7 point Likert scale from completely disagree=0, to completely agree=6
  1. Physical activity may cause pain
  2. Physical activity makes pain worse
  3. Physical activity might harm my tissues if I am hurting
  4. Physical activity should not be done if it increases pain
  5. Physical activities cannot be done if it makes pain worse
  score on a scale
    question 1 | 4.7 (1.5)
    question 2 | 3.6 (1.7)
    question 3 | 3.6 (1.3)
    question 4 | 5.1 (1.2)
    question 5 | 3.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Beliefs Questionnaire Score After VR Intervention Approximately 45 Minutes Later
Description: Pain beliefs questionnaire: 11 point Likert scale (0= strongly disagree, 10= strongly agree) on 5 pain beliefs questions. Some questions are positively worded so higher scores = more positive beliefs (#1, 4, 5). Some are negatively worded so higher scores = worse beliefs (#2, 3) question 1 - Pain is normal; without being able to feel pain you will not survive question 2 - Pain means something is wrong with your tissues question 3 - Pain always means you have to stop what you are doing question 4 - You can control how much pain you feel question 5 - Your brain decides if you feel pain, not your tissues
Time Frame: Baseline and immediately post intervention, intervention approximately 45 minutes of viewing Pain VR
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Middle School VR Students
Number analyzed (Participants) | 20
score on a scale
  question 1 | .35 (2.6)
  question 2 | .95 (3.1)
  question 3 | .45 (2.4)
  question 4 | .55 (2.7)
  question 5 | -.1 (2.6)
Statistical Analysis 1: Comparison: Middle School VR Students; Test type: Other — Paired samples pre-post t-test; p = .137, t-test, 2 sided

2. Primary Outcome: Change in Baseline Revised Neurophysiology of Pain Questionnaire to Post Intervention of VR, Approximately 45 Minutes Later
Description: 12 true false questions, higher scores of correct answers demonstrate higher pain knowledge. 12 points is highest score, 0 points is lowest score
Time Frame: Change in baseline score immediately post intervention, approximately 45 minutes after VR intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Middle School VR Students
Number analyzed (Participants) | 20
score on a scale | 1.45 (1.8)
Statistical Analysis 1: Comparison: Middle School VR Students; Test type: Other — Paired samples t-test (pre - post measure of group); p = .010, t-test, 2 sided

3. Primary Outcome: Change in Baseline Physical Activity Subscale of the Fear Avoidance Belief Questionnaire Scores to Post VR Viewing, Approximately 45 Minutes Later
Description: 7 point Likert scale (0= completely disagree, 6=completely agree), 5 questions (question 1-Physical activity may cause pain, question 2-Physical activity makes pain worse, question 3-Physical activity might harm my tissues if I am hurting, question 4-Physical activity should not be done if it increases pain, question 5-Physical activities cannot be done if it makes pain worse). The higher the score the higher the fear avoidance beliefs. Lowest score 0, highest score 30.
Time Frame: Change in baseline score immediately post intervention of viewing VR, approximately 45 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Middle School VR Students
Number analyzed (Participants) | 20
score on a scale
  question 1 | .2 (1.2)
  question 2 | -.05 (2.3)
  question 3 | .55 (2.0)
  question 4 | -1.0 (1.8)
  question 5 | -.35 (1.9)
Statistical Analysis 1: Comparison: Middle School VR Students; Test type: Other — Paired samples t-test (pre post measure of group); p = .591, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for from the start of Virtual reality during the entire educational session (approximately 45 minutes) and then after completion of the VR educational experience for 15 minutes while the completed the ending data collection. 1 hour total time.
Description: any episode of ill feeling while performing the VR or immediately (15 minutes) after performing VR
Arm/Group | Middle School VR Students
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT04470375/Prot_000.pdf
  • Informed Consent Form (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT04470375/ICF_001.pdf